CLINICAL TRIAL: NCT06674200
Title: A Retrospective Study Comparing the Incidence of Parastomal Hernia After Mesenteric Molding Suturing and Non-molding Suturing in Colostomy Surgery
Acronym: COMPARISON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Yueming Sun, Prof., The First Affiliated Hospital with Nanjing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMPARISON study
Record Dates: First submitted 2024-10-30; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer (CRC)
Keywords: Parastomal Hernia; Mesenteric Molding Suturing; Colostomy Surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regular (Active Comparator): The stoma surgery is performed using conventional non-molding suturing techniques. The specific steps include:
  Select an appropriate stoma site, typically within the rectus abdominis muscle. Perform routine suturing around the stoma without additional mesentery shaping. Form the stoma, ensuring a tight fit of the surrounding tissues.
  Interventions: Procedure: Mesenteric Molding Suturing Group
- Mesenteric Molding Suturing Group (Experimental): During the stoma surgery, the mesentery is shaped and sutured to enhance the support around the stoma and reduce the risk of hernia formation. The specific steps include:
  Select an appropriate stoma site, typically within the rectus abdominis muscle. Separate the mesentery around the stoma and shape it into a sturdy support structure.
  Use non-absorbable sutures to fix the shaped mesentery to the abdominal wall, forming a sturdy support structure.
  Form the stoma on the support structure, ensuring a tight fit of the surrounding tissues.
  Interventions: Procedure: Regular

INTERVENTIONS:
Procedure: Mesenteric Molding Suturing Group — During the stoma surgery, the mesentery is shaped and sutured to enhance the support around the stoma and reduce the risk of hernia formation. The specific steps include:
  Select an appropriate stoma site, typically within the rectus abdominis muscle. Separate the mesentery around the stoma and shape it into a sturdy support structure.
  Use non-absorbable sutures to fix the shaped mesentery to the abdominal wall, forming a sturdy support structure.
  Form the stoma on the support structure, ensuring a tight fit of the surrounding tissues.
  Arms: Regular
Procedure: Regular — The stoma surgery is performed using conventional non-molding suturing techniques. The specific steps include:
  Select an appropriate stoma site, typically within the rectus abdominis muscle. Perform routine suturing around the stoma without additional mesentery shaping. Form the stoma, ensuring a tight fit of the surrounding tissues.
  Arms: Mesenteric Molding Suturing Group

SUMMARY:
### Brief Summary

* Title**: A Retrospective Study Comparing the Incidence of Parastomal Hernia After Mesenteric Molding Suturing and Non-molding Suturing in Colostomy Surgery
* Background**:

Colostomy surgery is a common procedure for treating various gastrointestinal diseases, but it is associated with a high incidence of parastomal hernia (PSH), which can significantly affect patients' quality of life and increase healthcare costs. This study aims to compare the incidence of PSH within one year after colostomy surgery between patients who underwent mesenteric molding suturing and those who underwent non-molding suturing.

* Objectives**:

  * **Primary Objective**: To compare the incidence of PSH within one year postoperatively between the mesenteric molding suturing group and the non-molding suturing group.
  * **Secondary Objectives**: To evaluate the impact of the two suturing methods on stoma-related complications (such as stoma bleeding, stoma necrosis, and stoma prolapse), operative time, and time to stoma function recovery.
* Methods**:

  * **Design**: Retrospective cohort study.
  * **Participants**: Patients who underwent colostomy surgery.
  * **Interventions**: Mesenteric molding suturing vs. non-molding suturing.
  * **Data Collection**: Baseline data (age, gender, BMI, medical history) and follow-up data (incidence of PSH, stoma-related complications, operative time, and time to stoma function recovery) were collected from medical records.
  * **Statistical Analysis**: The primary outcome (incidence of PSH) will be analyzed using the Chi-square test or Fisher's exact test. Secondary outcomes will be analyzed using appropriate statistical methods (e.g., t-test, Mann-Whitney U test, ANOVA).
* Expected Outcomes**:

  - The study aims to provide evidence on the effectiveness of mesenteric molding suturing in reducing the incidence of PSH and improving postoperative outcomes in colostomy patients.
* Ethical Considerations**:

  * The study will adhere to the principles of the Declaration of Helsinki.
  * All data will be anonymized to protect patient confidentiality.
  * The study protocol will be approved by the local ethics committee.

This retrospective study will contribute valuable insights into the optimal surgical techniques for reducing the incidence of PSH in colostomy patients, ultimately improving their quality of life and reducing healthcare costs.

DETAILED DESCRIPTION:
* Detailed Description

  * Title A Retrospective Study Comparing the Incidence of Parastomal Hernia After Mesenteric Molding Suturing and Non-molding Suturing in Colostomy Surgery
  * Background Colostomy surgery is a common procedure used for the treatment of various gastrointestinal diseases, including rectal cancer, ulcerative colitis, and Crohn's disease. Despite its benefits, colostomy surgery is associated with a high incidence of postoperative complications, particularly parastomal hernia (PSH). PSH, defined as the formation of an abdominal wall hernia around the stoma, can occur in up to 50% of cases. PSH not only affects patients' quality of life but can also lead to pain, stoma dysfunction, and the need for reoperation, increasing medical costs and patient burden. Therefore, identifying effective strategies to prevent PSH is crucial.
  * Objectives

    * **Primary Objective**: To compare the incidence of parastomal hernia within one year after colostomy surgery between patients who underwent mesenteric molding suturing and those who underwent non-molding suturing.
    * **Secondary Objectives**:
    * To evaluate the impact of the two suturing methods on stoma-related complications such as stoma bleeding, stoma necrosis, and stoma prolapse.
    * To record the operative time and the time to stoma function recovery.
    * To assess changes in patients' quality of life.
  * Methods

    * **Design**: Retrospective cohort study.
    * **Setting**: The study will be conducted at [Hospital Name], a tertiary care center with a dedicated colorectal surgery unit.
    * **Participants**: Patients who underwent colostomy surgery between [Start Date] and [End Date].
    * **Inclusion Criteria**:
    * Age 18 years or older.
    * Underwent colostomy surgery.
    * Provided written informed consent.
    * Expected survival of more than one year.
    * No severe comorbidities such as heart, lung, liver, or kidney dysfunction.
    * **Exclusion Criteria**:
    * Pregnant or breastfeeding women.
    * History of major abdominal surgery that could affect the development of PSH.
    * Mental illness that impairs understanding of the study content and ability to give informed consent.
    * Patients receiving immunosuppressive therapy or chemotherapy.
  * Interventions

    * **Mesenteric Molding Suturing Group**:
    * During the stoma surgery, the mesentery is shaped and sutured to enhance the support around the stoma and reduce the risk of hernia formation. The specific steps include:

      1. Select an appropriate stoma site, typically within the rectus abdominis muscle.
      2. Separate the mesentery around the stoma and shape it into a sturdy support structure.
      3. Use non-absorbable sutures to fix the shaped mesentery to the abdominal wall, forming a sturdy support structure.
      4. Form the stoma on the support structure, ensuring a tight fit of the surrounding tissues.
    * **Non-molding Suturing Group**:
    * The stoma surgery is performed using conventional non-molding suturing techniques. The specific steps include:

      1. Select an appropriate stoma site, typically within the rectus abdominis muscle.
      2. Perform routine suturing around the stoma without additional mesentery shaping.
      3. Form the stoma, ensuring a tight fit of the surrounding tissues.
  * Data Collection - **Baseline Data**:

    * Patient demographic information: age, gender, BMI, etc.
    * Medical history: including surgical history and chronic disease history.
    * Laboratory tests: complete blood count, biochemical indicators, etc.
    * **Follow-up Data**:
    * **One Week Postoperatively**: Assess wound healing, record operative time, and time to stoma function recovery.
    * **One Month Postoperatively**: Evaluate stoma function and record complications such as stoma bleeding, stoma necrosis, and stoma prolapse.
    * **Six Months Postoperatively**: Repeat the above assessments and perform imaging studies (e.g., ultrasound or CT) to evaluate the incidence of PSH.
    * **One Year Postoperatively**: Repeat the above assessments and conduct the final statistical analysis of PSH incidence.
  * Statistical Analysis - **Primary Outcome Measure**: Incidence of PSH within one year postoperatively.

    - Compare the two groups using the Chi-square test or Fisher's exact test.
    * **Secondary Outcome Measures**:
    * Incidence of stoma-related complications such as stoma bleeding, stoma necrosis, and stoma prolapse: use the Chi-square test or Fisher's exact test.
    * Operative time and time to stoma function recovery: use the t-test or Mann-Whitney U test.
    * Quality of life assessment: use ANOVA or Kruskal-Wallis test.
    * **Multivariate Analysis**: Use Cox proportional hazards model to assess risk factors for PSH.
  * Ethical Considerations - The study will adhere to the principles of the Declaration of Helsinki.

    - All participants must provide written informed consent.

    - The study protocol must be approved by the local ethics committee.

    - Data will be anonymized to protect patient confidentiality.
  * Expected Outcomes - This study aims to provide scientific evidence for best practices in colostomy surgery, particularly in reducing PSH and other complications.

    - We expect to validate the effectiveness of mesenteric molding suturing in preventing PSH, offering more reliable surgical guidance for clinicians.
  * Study Limitations

    * **Open-label Design**: May introduce some bias, but it is difficult to achieve double-blinding given the nature of the surgical procedures.
    * **Long-term Follow-up**: May result in some dropouts, so measures will be taken to minimize the dropout rate.
    * **Sample Selection**: Potential selection bias, so strict inclusion and exclusion criteria will be applied.

By conducting this detailed retrospective study, we aim to provide robust evidence to guide clinical practice and improve the outcomes for patients undergoing colostomy surgery.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years or older. Patients requiring colostomy surgery. Ability to provide written informed consent. Expected survival of more than one year. No severe comorbidities such as heart, lung, liver, or kidney dysfunction.

Exclusion Criteria:

Pregnant or breastfeeding women. History of major abdominal surgery that could affect the development of PSH. Mental illness that impairs understanding of the study content and ability to give informed consent.

Patients receiving immunosuppressive therapy or chemotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11243 (Actual)
Dates: Start 2002-01-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Incidence of PSH within one year postoperatively | 1 year
  Incidence of PSH within one year postoperatively

SECONDARY OUTCOMES:
Incidence of stoma-related complications | 1 year
  stoma bleeding, stoma necrosis, and stoma prolapse: use the Chi-square test or Fisher's exact test.
Operative time and time to stoma function recovery | 1 year
  Operative time and time to stoma function recovery

IPD SHARING:
Plan to Share IPD: No